CLINICAL TRIAL: NCT02340845
Title: The Methods and Compositions for Treating / Preventing Various Types of Cancer Which Comprise Administered an Effective Amount of Glyco-Polypeptides, Such as Comosain, Bromelainases, Ananase, and a Mixture Thereof. By Way of (a) MMAPKinase (Major Mitogen Activiting Protein Kinase), (b) TPKinase (Tryosine Phosphorylation Kinase) Inhibitors Which Induce Cascade Production of Interleukin II B, 6, 8 & TNFs Through TCRs/ CD-2, TCRs/ CD-3 of WBC
Brief Title: Bromelain, Comosain as a New Drug for Treating and Preventing Various Types of Cancer in the Humans
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oeyama-Moto Cancer Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 116911
Record Dates: First submitted 2014-09-18; First posted 2015-01-19 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Cancer
Keywords: breast,colon, ovary, uterus, cervix, lung; Treatments
MeSH Terms: conditions — Neoplasms | interventions — Bromelains; comosain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bromalian 10 mg/kg/day (Active Comparator): The number of patients suffering from well-documented malignancies to be assigned to this group will be at least 30: with mixed types of carcinoma of breast, lung, colon, gastro-intestinal, ovarian, cervical, uterine, prostatic, bladder, hepatic, lymphoma, melanoma and so forth. These patients will be given Bromelain at 500 mg/day, divided into two doses of 250 mg/dose and taken with meals.
  Interventions: Biological: Bromelain and Comosain
- Bromalian 50mg/kg/day (Active Comparator): The number of patients suffering from well-documented malignancies with be at least 60: with mixed types of carcinoma of breast, lung, colon, gastro-intestinal, ovarian, cervical, uterine, prostatic, bladder, hepatic, lymphoma, melanoma and so forth. These patients will be given Bromelain at 2400 mg/day, divided into two doses of 1200 mg/dose and taken with meals.
  Interventions: Biological: Bromelain and Comosain

INTERVENTIONS:
Biological: Bromelain and Comosain — Treatment of solid tumors in advanced stage of lung, breast, colon, ovary, cervix, uterus, prostatic, and liver
  Other Names: Ananase, Comosalin, Bromelainase, Formosain, Formosalin

SUMMARY:
The Phase II randomized, two-armed clinical study will investigate the efficacy of high dose versus low dose Bromelain (Comosain) in human subjects diagnosed with advanced late stage cancers. The study subjects will be randomly assigned to each group by a coin toss. Bromelain (Comosain) extract, derived from the stem and fruit of Ananas Comosus will be administered orally each day.

DETAILED DESCRIPTION:
1. Patient Eligibility and Selection

   Patients suffering from late stage breast, lung, colon, cervical, ovarian, and uterine cancers in stages III and IV, with tissue proof of well-documented malignancies, whether by tissue biopsies and/or laparatomy or thoracotomy and have not been helped by conventional radiation therapy and/or chemotherapies are eligible for this study. Additionally the following conditions must be met:
   1. Patient's age is between 18 and 85 years.
   2. Patient is not taking anticoagulants or on antiplatelet therapy.
   3. Patient does not have a history of abdominal fistula, gastroenteral perforation, peptic ulcer diseases, or intra-abdominal abscess within 6 months prior to study enrollment.
   4. Patient has not had major surgery within 4 weeks prior to study enrollment. Patients who have not recovered from adverse events due to surgery performed more than 4 weeks earlier are not eligible for this study.
   5. Patient does not currently have uncontrolled hypertension, diabetes, or clinically significant cardiac arrhythmia.
   6. Patient does not have an allergic reaction to Bromelain or pineapple-containing products.
   7. Female patients should not be pregnant or breastfeeding.
   8. Patient's platelet counts must be greater than 100,000/mL.
   9. Patient's hemoglobin must be greater than 9.0 g/dL.
   10. Patient does not have significant abnormal hepatic and/or renal function.
   11. Patient's tumors are measurable; between 0.2 - 10 cm in size and number between 1 - 15. All measurable tumors that have spread to the bones, liver, lung, kidney, and abdomen will be included in the data analysis.

   Patients with following conditions will be excluded from the study:
   1. Hemoglobulin less than 9 g/dL and WBC less than 4.0 k/µL.
   2. Platelet count less than 100,000/µL.
   3. INR greater than 1.5
   4. Patient currently taking therapeutic doses of warfarin or anti anti-platelet agents.
   5. Patient has a history of abdominal fistula, gastrointestinal perforation, peptic ulcer disease, or intra-abdominal abscess within 6 months prior to study enrollment.
   6. Patient currently has uncontrolled hypertension, diabetes, or clinically significant cardiac arrhythmia.
   7. Patient who had major surgery performed within 4 weeks prior to entering the study; and patients who have not recovered from adverse events due to surgery performed more than 4 weeks earlier.
   8. Patient with a history of allergic reaction to Bromelain or pineapple-containing products.
   9. Female patients who are pregnant or breastfeeding.
   10. Patient with tumors that are widely spread in the chest and abdomen that cannot be measured by CT scan.

   Patients who are eligible for this study will be randomly assigned to either the low dose group or the high dose group by a coin toss. Each study subject will be assigned a patient number for the purpose of this study.
2. Drug Dosage and Schedule

   High Dose Group-The oral dose of Bromelain (50 mg/kg/day) is extrapolated from in vivo animal studies, and determined to be safe by a Safety study on healthy human subjects (see Section VII-A). For this clinical investigation, the High Dose group will be given Bromelain at 50 mg/kg/day, to a maximum of 2400 mg/day (divided into 2 doses/day of 1200 mg/dose)

   Low Dose Group - Low Dose group will be given 10 mg/kg/day, to a maximum of 500 mg/day (divided into 2 doses/day of 250 mg/dose).

   The number of patients suffering from well-documented malignancies to be assigned to this group will be at least 30: with the combination of mixed types carcinoma of breast, lung, colon, gastro-intestinal, ovarian, cervical, uterine, prostatic, hepatic, bladder, lymphoma, melanoma, and so forth. These patients will be given Bromelain at 500 mg/day, divided into two doses of 250 mg/dose and taken with meals.

   High Dose Group - The dose will be at 50 mg/kg/day, The number of patients suffering from well-documented malignancies with be at least 60: with the combination of mixed types carcinoma of breast, lung, colon, gastro-intestinal, ovarian, cervical, uterine, prostatic, hepatic, bladder, lymphoma, melanoma, and so forth. These patients will be given Bromelain at 2400 mg/day, divided into two doses of 1200 mg/dose and taken with meals.
3. Duration and Route of Administration Study subjects will be provided with Bromelain for oral administration. The containers will be clearly labeled (see Section V-E). Bromelain will be taken orally twice daily with meals. On their biweekly visits to the Doctor's Office, the Study patients will be provided with enough doses for two weeks. The study patients are required to keep a journal of the daily doses they take and any side effects they experience.

The study patients will be evaluated using blood tests and CT scans at six months for signs of disease progression. If the disease did not progress, then treatment will continue and the patient will be evaluated every six months thereafter until the investigator determines otherwise. If the disease did progress, then the patient will be taken off the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from late stage breast, lung, colon, cervical, ovarian, and uterine cancers in stages III and IV, with tissue proof of well-documented malignancies, whether by tissue biopsies and/or laparatomy or thoracotomy and have not been helped by conventional radiation therapy and/or chemotherapies are eligible for this study. Additionally the following conditions must be met:

  1. Patient's age is between 18 and 85 years.
  2. Patient is not taking anticoagulants or on antiplatelet therapy.
  3. Patient does not have a history of abdominal fistula, gastroenteral perforation, peptic ulcer diseases, or intra-abdominal abscess within 6 months prior to study enrollment.
  4. Patient has not had major surgery within 4 weeks prior to study enrollment. Patients who have not recovered from adverse events due to surgery performed more than 4 weeks earlier are not eligible for this study.
  5. Patient does not currently have uncontrolled hypertension, diabetes, or clinically significant cardiac arrhythmia.
  6. Patient does not have an allergic reaction to Bromelain or pineapple-containing products.
  7. Female patients should not be pregnant or breastfeeding.
  8. Patient's platelet counts must be greater than 100,000/mL.
  9. Patient's hemoglobin must be greater than 9.0 g/dL.
  10. Patient does not have significant abnormal hepatic and/or renal function.
  11. Patient's tumors are measurable; between 0.2 - 10 cm in size and number between 1 - 15. All measurable tumors that have spread to the bones, liver, lung, kidney, and abdomen will be included in the data analysis.

Exclusion Criteria:

* Patients with following conditions will be excluded from the study:

  1. Hemoglobulin less than 9 g/dL and WBC less than 4.0 k/µL.
  2. Platelet count less than 100,000/µL.
  3. INR greater than 1.5
  4. Patient currently taking therapeutic doses of warfarin or anti anti-platelet agents.
  5. Patient has a history of abdominal fistula, gastrointestinal perforation, peptic ulcer disease, or intra-abdominal abscess within 6 months prior to study enrollment.
  6. Patient currently has uncontrolled hypertension, diabetes, or clinically significant cardiac arrhythmia.
  7. Patient who had major surgery performed within 4 weeks prior to entering the study; and patients who have not recovered from adverse events due to surgery performed more than 4 weeks earlier.
  8. Patient with a history of allergic reaction to Bromelain or pineapple-containing products.
  9. Female patients who are pregnant or breastfeeding.
  10. Patient with tumors that are widely spread in the chest and abdomen that cannot be measured by CT scan.

Patients who are eligible for this study will be randomly assigned to either the low dose group or the high dose group by a coin toss. Each study subject will be assigned a patient number for the purpose of this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Using NCI standard measurement to measure primary target lesion size of various types of cancer pstients | 24 weeks
  Measurement of the size of tumor lesion in centimeters and shrinking of regional lymphnodes

SECONDARY OUTCOMES:
Using NCI standard measurement to measure non-target lesion (tumor markers) value in various types of cancer patients | 24 weeks
  Measurement of the non-target lesions (tumor markers) values decrease or increase by laboratory tests

OTHER OUTCOMES:
Using NCI standard to measure serious and non-serious outcomes in toxicity in various types of cancer patients | 24 weeks
  Using standard serious and non-serious toxicity measurement in hematology, hepato-reno systems in cancer patients

CONTACTS AND LOCATIONS:
Overall Officials: Benedict Liao, M.D., Principal Investigator — OeyamaMoto Cancer research Foundation
Locations (1):
- OeyamaMoto Cancer Research Foundation, West Covina, California, United States